CLINICAL TRIAL: NCT00696059
Title: Can Bone Erosions Heal in Adalimumab (Humira) Treated Rheumatoid Arthritis Patients. An Imaging Study Using Computed Tomography and Magnetic Resonance Imaging.
Brief Title: Humira in Rheumatoid Arthritis - Do Bone Erosions Heal?
Acronym: HURRAH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Mikkel Østergaard, Department of Rheumatology, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM 04-20
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Rheumatoid Arthritis; Arthritis; Joint Diseases
Keywords: Rheumatoid arthritis; Computed tomography; Magnetic resonance imaging; Radiography; Tumor necrosis factor alpha antagonists
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Joint Diseases | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Open-label, one arm only. All patients receiving active drug according to recommendations (adalimumab (Humira) 40 mg subcutaneously every other week).
  Interventions: Drug: Adalimumab (Humira)

INTERVENTIONS:
Drug: Adalimumab (Humira) — Adalimumab (Humira) 40 mg subcutaneously every other week
  Other Names: Humira

SUMMARY:
Studies on tumor necrosis factor alpha antagonist (anti-TNF) therapy in rheumatoid arthritis (RA) patients have found that erosive damage may "heal" in some RA patients treated with anti-TNF. Repeated examinations of adalimumab (Humira) treated RA patients, using computed tomography (CT), magnetic resonance imaging (MRI), ultrasonography (US) and radiography will allow detailed assessment of the extent of bone repair/healing during adalimumab (Humira) therapy.

DETAILED DESCRIPTION:
Studies on tumor necrosis factor alpha antagonist (anti-TNF) therapy in rheumatoid arthritis (RA) patients have found that radiographic erosions scores decreased in some patients. This suggests that erosive damage may "heal" in some RA patients treated with anti-TNF. However, it is not clarified whether the reduced scores are caused by technical issues as observer variation and image acquisition differences. Furthermore, radiography of erosions is a 2D representation of a 3D pathology and therefore not ideal for visualizing healing, if present. Verification of erosion healing under anti-TNF therapy with adalimumab (Humira) by optimal imaging methods, would markedly influence our perception of the effect and potential of adalimumab (Humira) for modifying structural joint damage in RA. Magnetic Resonance Imaging (MRI), allowing high-resolution 3D visualization of bone damage as well as the inflammatory activity in the bone (bone marrow edema/osteitis), is more sensitive for visualization of bone erosions than radiography. Computed Tomography (CT) is a 3D radiographic imaging technique, which is not suited for assessment of inflammation, but can be considered a reference method for assessment of bone damage, due to its direct 3D visualization of calcified tissue. Internationally recommended MRI scoring systems as well as methods for estimation of erosion volumes have been developed, with participation by our research group. Ultrasonography (US), even though less validated, is more sensitive than radiography and comparable to MRI in detecting bone erosions in RA joints. Additionally, US provides visualisation of soft tissue changes and synovitis, using gray-scale and Doppler US.

Repeated MRI, CT, US and radiographic examinations of RA joints with mild to moderate radiographic damage under adalimumab (Humira) therapy will allow detailed assessment of the extent of bone repair/healing during adalimumab (Humira) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis according to the American College of Rheumatology 1987 criteria
* Moderate or severely active RA, defined as a DAS28(CRP)> 3.2
* Moderate radiographic structural joint damage, defined as Larsen grade 2-3, in ≥ 2 wrist and/or MCP joints
* No previous biological therapy
* Clinical indication for biological therapy, according to the treating physician
* Treatment with methotrexate and folic acid for at least 4 weeks prior to inclusion
* No history of tuberculosis, and no signs of tuberculosis at chest radiograph or Mantoux test.
* No contra-indications for TNF-alpha antagonist treatment
* Co-operability of the patient, including that the patient is willing and able to comply with the treatment and scheduled follow-up visits and examinations
* Oral and signed informed consent by the patient

Exclusion Criteria:

* Acute infection, and known chronic viral infection such as HIV or hepatitis B and C
* Other DMARDs than methotrexate within last 4 weeks before inclusion
* Intramuscular or intraarticular glucocorticoids within last 4 weeks before inclusion
* Oral treatment with prednisolone >10 mg per day
* Malignant lymphoma and other malignant disease
* Other serious concomitant diseases (uncontrolled/severe kidney, liver, haematological, gastrointestinal, endocrine, cardiovascular, pulmonary, neurological or cerebral disease (including demyelinating disease))
* Pregnancy and lactation. Patients must use safe anti-conception during the treatment.
* Development of SLE-like disease. Occurrence of positive ANA and/or anti-DNA antibodies without clinical symptoms is not considered a contra-indication.
* Contra-indications for MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
By means of computed tomography and magnetic resonance imaging to investigate if repair of bone erosion occurs in rheumatoid arthritis joints during adalimumab (Humira) therapy | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Østergaard, Professor, Principal Investigator — Department of Rheumatology, Hvidovre University Hospital; Uffe Møller Døhn, M.D, Study Chair — Department of Rheumatology, Hvidovre University Hospital
Locations (5):
- Denmark (5):
  - Department of Rheumatology, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Rheumatology, Bispebjerg University Hospital, Copenhagen
  - Department of Rheumatology, Gentofte University Hospital, Hellerup
  - Department of Rheumatology, Herlev University Hospital, Herlev
  - Department of Rheumatology, Hvidovre University Hospital, Hvidovre

REFERENCES:
- [Derived] Krabbe S, Bolce R, Brahe CH, Dohn UM, Ejbjerg BJ, Hetland ML, Sasso EH, Chernoff D, Hansen MS, Knudsen LS, Hansen A, Madsen OR, Hasselquist M, Moller J, Ostergaard M. Investigation of a multi-biomarker disease activity score in rheumatoid arthritis by comparison with magnetic resonance imaging, computed tomography, ultrasonography, and radiography parameters of inflammation and damage. Scand J Rheumatol. 2017 Sep;46(5):353-358. doi: 10.1080/03009742.2016.1211315. Epub 2016 Sep 28. PMID 27682742